CLINICAL TRIAL: NCT01129947
Title: The Use of DHEA in Women With Premature Ovarian Failure
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: very poor patient recruitement
Sponsor: Virginia Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Fady I. Sharara, M.D, Medical Director, Virginia Center for Reproductive Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCRM4
Record Dates: First submitted 2010-05-23; First posted 2010-05-25 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DHEA (Experimental)
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: DHEA — DHEA 25 mg tid

SUMMARY:
DHEA supplementation has been used in women with infertility and diminished ovarian reserve. There is a small report in 5 women with POF that benefited from the use of DHEA over several months. The investigators aim to evaluate further the use of DHEA in women with Premature ovarian failure (POF).

ELIGIBILITY:
Inclusion Criteria:

* women with POF

Exclusion Criteria:

* women without ovaries

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The Use of DHEA in Women With Premature Ovarian Failure | 3 years
  The following outcomes will be evaluated: FSH, AMH, estradiol, ovarian volume, antral follicle count, pregnancy in women seeking to conceive

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Center for Reproductive Medicine, Reston, Virginia, United States

REFERENCES:
- [Background] Mamas L, Mamas E. Dehydroepiandrosterone supplementation in assisted reproduction: rationale and results. Curr Opin Obstet Gynecol. 2009 Aug;21(4):306-8. doi: 10.1097/gco.0b013e32832e0785. PMID 19610174